CLINICAL TRIAL: NCT00624936
Title: Phase I Study of Vidaza and Velcade (Bortezomib) in Acute Myeloid Leukemia
Brief Title: Azacytidine and Bortezomib in Treating Patients With Relapsed or Refractory Acute Myeloid Leukemia or Myelodysplastic Syndromes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry); Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-07095; NCI-2011-03146 (Registry Identifier: Clinical Trial Reporting Program (CTRP))
Record Dates: First submitted 2008-02-27; First posted 2008-02-28 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Leukemia; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms
Keywords: adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); recurrent adult acute myeloid leukemia; myelodysplastic/myeloproliferative neoplasm, unclassifiable; myelodysplastic syndromes; secondary acute myeloid leukemia
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Congenital Abnormalities; Leukemia, Myeloid, Acute; Myeloproliferative Disorders | interventions — Azacitidine; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vidaza and Velcade (Experimental): Vidaza 75mg/m2 IV over 30 min daily on days 1-7 This dose is the same for all dose levels. Velcade will be given immediately after Vidaza is completed at one of the following dose levels: 1, 2, 3, 4
  Interventions: Drug: Vidaza; Drug: Velcade

INTERVENTIONS:
Drug: Vidaza — Vidaza 75mg/m2 IV over 30min daily on days 1-7. This dose is the same for all dose levels.
  Other Names: Azacitidina; Azacitidinum; Azacytidine; Mylosar
Drug: Velcade — Dose level 1 Velcade 0.7mg/m2 IVP on days 2 and 5 Dose level 2 Velcade 0.7mg/m2 IVP on days 2, 5, 9, 12 Dose level 3 Velcade 1.0 mg/m2 IVP on days 2, 5, 9, 12 Dose level 4 Velcade 1.3 mg/m2 IVP on days 2, 5, 9, 12
  Other Names: Bortezomib

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as azacytidine work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Bortezomib may stop the growth of cancer cells by blocking blood flow to the cancer and by blocking some of the enzymes needed for cell growth. Giving azacytidine together with bortezomib may kill more cancer cells.

PURPOSE: This phase I trial is studying the side effects and best dose of bortezomib when giving together with azacytidine in treating patients with relapsed or refractory acute myeloid leukemia or myelodysplastic syndromes.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the maximum tolerated dose (MTD) bortezomib in combination with Azacytidine in patients with relapsed/refractory acute myeloid leukemia (AML) and myelodysplastic syndromes (MDS).
* To define the specific toxicities and the dose limiting toxicity (DLT) of Azacytidine plus bortezomib combination.

Secondary

* To determine the overall response rate (ORR).
* To determine the rate of complete remission (CR) of Azacytidine plus bortezomib in relapsed/refractory AML and MDS.
* To correlate the biological activity of Azacytidine as demethylating agent (changes in target gene methylation and gene expression, DNMT1 protein expression, global methylation) with clinical endpoints and plasma pharmacokinetics of azacytidine.
* To characterize the biological activity of bortezomib as a potential demethylating agent.
* To correlate intracellular concentration of azacytidine-triphosphate with global DNA methylation and other biological endpoints as well as clinical response.
* To explore the biologic role of microRNAs in determining clinical response to the azacytidine plus bortezomib combination and achievement of the other pharmacodynamic endpoints.

OUTLINE: This is a dose-escalation study of bortezomib.

Patients receive azacytidine IV over 30 minutes on days 1-7 and bortezomib IV on days 2 and 5 or on days 2, 5, and 9 or on days 2, 5, 9, and 12. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of bortezomib and tipifarnib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

After completion of study treatment, patients are followed for at least 30 days.

ELIGIBILITY:
Inclusion criteria:

* Patients must be >18 with relapsed or refractory acute myeloid leukemia (AML) and high risk (by IPSS scoring) Myelodysplastic Syndromes (MDS)
* Patients with secondary AML or therapy related disease (t-AML) are eligible If decitabine or Vidaza was a prior treatment for MDS or AML patient is eligible.Prior Velcade is also permitted.
* ECOG performance status 0-2
* Life expectancy > 6 months for patients with a co-morbid medical illness
* Total bilirubin < 2.0mg/dL
* AST/ALT < 2.5 times upper limit of normal (ULN)
* Creatinine < 2.0 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception prior to and during study treatment
* Ability to understand and willingness to sign the written informed consent document
* Active infection is allowed provided it is under control

Exclusion criteria:

* History of allergic reactions attributed to compounds of similar chemical or biologic composition to azacytidine or bortezomib that are not easily managed
* Hypersensitivity to bortezomib, boron, or mannitol
* Uncontrolled intercurrent illness including, but not limited to:

  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Serious cardiac arrhythmia
  * Psychiatric illness/social situations that would limit compliance with study
* Myocardial infarction within 6 months prior to enrollment
* New York Heart Association (NYHA) Class III or IV congestive heart failure
* Uncontrolled angina
* Severe uncontrolled ventricular arrhythmia
* Electrocardiographic evidence of acute ischemia
* Active conduction system abnormalities
* ECG abnormality that is medically relevant
* Psychiatric conditions that prevent compliance with protocol or consent.
* Pre-existing neuropathy grade 2 or higher or other serious neurologic toxicity that would significantly increase risk of complications from bevacizumab therapy
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study
* Diagnosis or treatment for another malignancy within 3 years of enrollment, with the exception of any of the following:

  * Complete resected basal cell carcinoma
  * Squamous cell carcinoma of the skin
  * Any in situ malignancy
  * Low-risk prostate cancer after curative therapy

PRIOR CONCURRENT THERAPY:

* Prior decitabine or azacytidine for MDS or AML is allowed
* Prior bortezomib allowed
* More than 2 weeks since prior chemotherapy or radiotherapy (6 weeks for nitrosoureas or mitomycin C)
* More than 14 days since prior and no concurrent investigational agents
* No concurrent combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2008-04 (Actual); Primary Completion 2009-12 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of bortezomib in combination with azacytidine | Up to 1 year
  Determine the maximum tolerated dose (MTD) of Velcade (bortezomib, PS-341) in combination with Vidaza in patients with relapsed/refractory acute myeloid leukemia (AML) and Myelodysplastic Syndrome (MDS)
Overall response rate | Up to 1 year
  Determine the overall response rate (ORR)

SECONDARY OUTCOMES:
Rate of complete remission | Up to 1 year
  Determine the rate of complete remission (CR) of Vidaza plus Velcade in relapsed/refractory AML and MDS
Biological activity of azacytidine and bortezomib as demethylating agents | Up to 1 year
  Correlate the biological activity of Vidaza as demethylating agent (changes in target gene methylation and gene expression, DNMT1 protein expression, global methylation) with clinical endpoints and plasma pharmacokinetics of Vidaza
Correlation of intracellular concentration of azacytidine-triphosphate with global DNA methylation and other biological endpoints as well as clinical response | Up to 1 year
  Characterize the biological activity of Velcade as a potential demethylating
Biologic role of microRNAs in determining clinical response to study drugs | Up to 1 year
  Correlate intracellular concentration of Vidaza-triphosphate with global DNA methylation and other biological endpoints as well as clinical response
Achievement of other pharmacodynamic endpoints | Up to 1 year
  Explore the biologic role of microRNAs in determining clinical response to the Vidaza plus Velcade combination and achievement of the other pharmacodynamic endpoints.

CONTACTS AND LOCATIONS:
Overall Officials: William G. Blum, MD, Principal Investigator — Ohio State University; Guido Marcucci, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- See also: Jamesline — http://cancer@osu.edu